CLINICAL TRIAL: NCT04540601
Title: Antiresorptive Drug Continuation Compared With Drug Holiday in Cancer Patients Needing Tooth Extraction - A Randomized Clinical Trial
Brief Title: Antiresorptive Drug Continuation Compared With Drug Holiday in Cancer Patients Needing Tooth Extraction
Acronym: DrugHoliday
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Department of Oral and Maxillofacial Surgery, Copenhagen University Hospital (Unknown)
Responsible Party: Principal Investigator, Camilla Ottesen, DDS, PhD fellow, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-18007990
Record Dates: First submitted 2020-08-24; First posted 2020-09-07 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Osteonecrosis Due to Drugs, Jaw

STUDY DESIGN:
Intervention Model Description: This trial is designed as an investigator-initiated, parallel-group, randomized, clinical, single-blinded, trial investigating no antiresorptive drug holiday starting before tooth extraction with primary closure versus antiresorptive drug holiday starting before tooth extraction with primary closure in cancer patients
Who Masked: Investigator, Outcomes Assessor
Masking Description: The allocation of the patients is not known to the clinical investigator, the surgeon or the outcome assessor but to the patient's oncologic doctor and nurse, who are in charge of drug delivery, and a supervisor (Klaus Gotfredsen) not involved in any registrations or surgeries.
  The participating patients will not be blinded. The patients do know which group they are randomized to and therefore do know if they are treated with or without drug holiday during the trial period (1+3 months). The patients are carefully instructed not to reveal which group they belong during the trial to the assessor.
  Klaus Gotfredsen will make sure that the patients randomized to the intervention group will continue their antiresorptive therapy and the patients randomized to the control group will be treated with drug holiday this in close collaboration with the oncological departments. The medicine will be giving to the patient by the department's nurse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cancer patients, randomized A (Active Comparator): Patients in high-dose antiresorptives with bone metastases
  Interventions: Other: Continuation of antiresorptives in relation to tooth extraction (surgical tooth removal)
- Cancer patients, randomized B (No Intervention): Drug Holiday as standard operation procedure

INTERVENTIONS:
Other: Continuation of antiresorptives in relation to tooth extraction (surgical tooth removal) — We want to investigate the importance of an antiresorptive drug holiday (bisphosphonate, denosumab) in relation to tooth extraction. The experimental intervention in this trial is drug continuation starting before tooth extraction with primary closure.
  We simply ask the participating cancer patients to continue their high dose antiresorptive treatment for 4 months (intervention-period: 1 month pre-operative, 3 months post-operative) instead of taking a drug holiday.
  Arms: Cancer patients, randomized A

SUMMARY:
The aim of this trial is to evaluate high-dose antiresorptive drug holiday related to tooth extraction with primary mucosal closure (surgical extraction) including how a drug holiday affects the health related quality of life.

Research question: Does a drug holiday have any influence on health related quality of life or the incidence of developing osteonecrosis of the jaw after surgical tooth extraction? The investigators hypothesize that a drug holiday 1 month before to 3 months after surgical tooth extraction in cancer patients do not influence the development of osteonecrosis of the jaw and may even affect the health related quality of life negatively.

DETAILED DESCRIPTION:
Osteonecrosis of the jaw is a known adverse reaction to antiresorptive medication, including bisphosphonate and denosumab. The globally accepted term is Medication-Related Osteonecrosis of the Jaws (MRONJ). Since 2003 there has been a worldwide focus at medication-related osteonecrosis, even though there still exist several of unanswered questions - one of them is the effect of a drug holiday in relation to tooth extraction. A drug holiday is a temporary discontinuation of a drug and has been suggested among risk reduction strategies in the literature. It is still unknown whether a drug holiday plays a significant role in relation to tooth extraction for the development of osteonecrosis. The investigators want to investigate the importance of an antiresorptive drug holiday (bisphosphonate, denosumab) in relation to tooth extraction.

The aim of this trial is therefore to clarify the meaning of high-dose antiresorptive drug holiday related to tooth extraction with primary mucosal closure in cancer patients and reveal how a drug holiday affects the health related quality of life. A continuation of the patients' antiresorptive treatment can possibly lead to increased risk of osteonecrosis of the jaw, but with the operation procedure with primary closure it is unlikely. It is beneficial for the cancer patients to continue the high dose antiresorptive therapy because a drug holiday is a stop in their anti-cancer treatment with risk of increased pain as well as unwanted skeletal events to occur, and potentially progress of metastases to follow.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the trial must comply with all of the following at randomization:
* Patients aged 18 years or older.
* Patients with malignant disease (breast or prostate cancer, multiple myeloma) and metastases to the skeleton.
* Patients present high dose/intravenous antiresorptive therapy for at least 1 month.
* Patients who need tooth extraction. Indications for extraction include root fracture, endodontic failure, severe periodontal disease, non-restorable caries and teeth with a poor prognosis or at high risk of infection, complications.
* Patients who have an ECOG (Eastern Cooperative Oncology Group) score < 2 (30). Definition of ECOG 0. Fully active, able to carry on all pre-disease performance without restriction.

  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g., light house work, office work.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of walking hours.
  3. Capable of only limited selfcare, confined to bed or chair more than 50% of walking hours.
  4. Completely disabled. Cannot carry on selfcare. Totally confined to bed or chair.
* Signed informed content.

Exclusion Criteria:

* Patients must not have received radiation therapy to the jaws.
* Patients must not have exposed bone, or signs of non-exposed bone.
* Patients previous diagnosed with ONJ.
* Patients who are unable to cooperate or too ill to complete the experiment.
* Lack of signed informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Development of osteonecrosis of the jaw (ONJ) or incomplete healing at 3 months follow-up | 3 months follow-up
  The outcome assessor has 3 options for registration related to ONJ occurrence:
  * Complete healing = mucosal covering = no sign of ONJ, defined as complete wound healing; Intact mucosa, that is total mucosal covering over the tooth extraction area.
  * Incomplete healing = presence of fibrin covering partly or over all mucosal operation area; Defined as the presence of fibrin at the surface of the operation area, thus still being a wound.
  * ONJ present, defined according to the AAOMS position paper 2014 (4), all three items have to be present:
    1. Current or previous treatment with antiresorptive agents.
    2. Exposed bone or bone that can be probed through an extraoral or intraoral fistula that has persisted for longer than 8 weeks.
    3. No history of radiation therapy to the jaws or obvious metastatic disease to the jaws.
EQ-5D-5L: Change in patients health related quality of life from allocation/enrollment | The patient will be asked to fulfill the EQ-5D-5L at allocation/enrollment and again at 1, 3 and 6 months follow-up.
  The patients are given the EQ-5D-5L questionnaire. The 5-level EQ-5D version (EQ-%D-5L) was introduced by the EuroQol Group in 2009 and consists of two pages: the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, serve problems and extreme problems. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The Danish dataset (SPSS syntax crosswalk values EQ-5D-5L Denmark) will be used to analyze patients´ responses.

SECONDARY OUTCOMES:
Pain from the jaw | This is asked prior to tooth extraction (time 0), at suture removal (time 10-14 days), at 1-month follow-up and at 3 and 6 months follow-up and is registered in the datasheet.
  Pain from the jaw is registered by a Visual Analogue Scale (VAS). The investigator will give the patient a paper with a VAS, see attached appendix 3, and ask following question: "On a scale from 0 to 10, where 0 is no pain and 10 is the worst thinkable pain, mark at the scale how much pain you feel from your jaw at tooth operation site".
Incidence of unwanted skeletal events | Incidence (number of) unwanted skeletal events during the period and is registered at 3 and 6 months follow-up.
  The patient is giving a simple questionnaire, where they have to answer yes or no to following question: "Have you visited your own doctor or been hospitalized because of fractures or other skeletal complications during this trial period - yes or no. If yes, please write why." See attached appendix 4: Skeletal-related event questionnaire
Progression of cancer disease | The patient will be weighted at baseline, time of tooth removal, 1 month follow-up, 3 and 6 months follow-up visit.
  The tumor-evaluation will be done by the oncologic doctor in due to their departments routine.

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen, Copenhagen Ø
  - University of Copenhagen, Department of Odontology, Copenhagen, Nørrebro

IPD SHARING:
Plan to Share IPD: No